CLINICAL TRIAL: NCT03325426
Title: ACtivity Trackers to ImproVe Blood Pressure: a Pilot Study
Brief Title: Activity Trackers for Improving BP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 16-18605
Record Dates: First submitted 2017-10-25; First posted 2017-10-30 (Actual); Results first posted 2022-07-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Hypertension; Cardiovascular Risk Factor; Physical Activity; Chronic Kidney Diseases
MeSH Terms: conditions — Hypertension; Motor Activity; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Usual care (No Intervention): No physical activity tracker or feedback x 6 months, then crossover to physical activity tracker x 6 months
- Physical activity tracker (Experimental): Physical activity tracker x 12 months (6 months with study feedback and 6 months without)
  Interventions: Device: FitBit

INTERVENTIONS:
Device: FitBit — Daily use of physical activity tracker coupled with biweekly provider telemonitoring and feedback for 6 months and then additionally without feedback for an additional 6 months
  Other Names: physical activity tracker
  Arms: Physical activity tracker

SUMMARY:
The study aims to determine if use of physical activity trackers coupled with provider feedback will increase awareness of young adults of their physical fitness and improve blood pressure levels. The goal of this pilot study is feasibility, with a secondary goal of examining potential effect sizes for planning purposes for a larger randomized controlled trial.

DETAILED DESCRIPTION:
Increasing physical activity levels may improve cardiovascular health and BP levels in young individuals, especially if such strategies promote healthy lifestyles. Physical activity is currently recommended for adults CV health, but physical activity levels are known to be low in populations with diabetes or chronic kidney disease. One prior study of the use of pedometers (not associated with wireless technology or provider feedback) in children with CKD did not significantly improve physical activity levels. Supervised walking appeared to provide some benefit in individuals with type II diabetes, but overall compliance was poor. Interview of adolescents and young adults with chronic illnesses has shown preference for the use of electronic devices and online tools for disease management.Thus, use of sophisticated electronic devices such as FitBits© (wireless pedometers worn on the wrist that sync with cell phones) may improve disease control by engaging young patients in self-monitoring of their own health and lifestyle behaviors. This pilot study aims to determine if use of FitBits© coupled with provider feedback will increase awareness of young adults of their physical fitness and improve blood pressure levels.

ELIGIBILITY:
Inclusion Criteria:

* ages 8-30 receiving anti-hypertensive therapy at the time of recruitment.
* diabetes, non-dialysis requiring chronic kidney disease, kidney transplant, or other etiologies of hypertension
* have phones compatible for wireless device (FitBits©) data transmission

Exclusion Criteria:

* history of decompensated congestive heart failure
* pregnant
* cognitive impairment
* unable to perform physical activity
* BP >180/110 mm Hg
* prisoners
* contraindication to use or wear of home activity tracker (such as allergy to activity tracker band)
* presence of any co-morbidity that would preclude physical activity
* actively using physical activity tracking devices prior to the study will be excluded.

Ages: 8 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Ku, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen DL, Huan Y, Townsend RR. Home blood pressure monitoring in CKD. Am J Kidney Dis. 2014 May;63(5):835-42. doi: 10.1053/j.ajkd.2013.12.015. Epub 2014 Feb 12. PMID 24529535
- [Background] Logan AG, McIsaac WJ, Tisler A, Irvine MJ, Saunders A, Dunai A, Rizo CA, Feig DS, Hamill M, Trudel M, Cafazzo JA. Mobile phone-based remote patient monitoring system for management of hypertension in diabetic patients. Am J Hypertens. 2007 Sep;20(9):942-8. doi: 10.1016/j.amjhyper.2007.03.020. PMID 17765133
- [Background] Agarwal R, Bills JE, Hecht TJ, Light RP. Role of home blood pressure monitoring in overcoming therapeutic inertia and improving hypertension control: a systematic review and meta-analysis. Hypertension. 2011 Jan;57(1):29-38. doi: 10.1161/HYPERTENSIONAHA.110.160911. Epub 2010 Nov 29. PMID 21115879
- [Background] Uhlig K, Balk EM, Patel K, Ip S, Kitsios GD, Obadan NO, Haynes SM, Stefan M, Rao M, Kong Win Chang L, Gaylor J, Iovin RC. Self-Measured Blood Pressure Monitoring: Comparative Effectiveness [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2012 Jan. Report No.: 12-EHC002-EF. Available from http://www.ncbi.nlm.nih.gov/books/NBK84604/ PMID 22439158
- [Background] Akber A, Portale AA, Johansen KL. Pedometer-assessed physical activity in children and young adults with CKD. Clin J Am Soc Nephrol. 2012 May;7(5):720-6. doi: 10.2215/CJN.06330611. Epub 2012 Mar 15. PMID 22422539
- [Background] Mohammed J, Deda L, Clarson CL, Stein RI, Cuerden MS, Mahmud FH. Assessment of habitual physical activity in adolescents with type 1 diabetes. Can J Diabetes. 2014 Aug;38(4):250-5. doi: 10.1016/j.jcjd.2014.05.010. PMID 25092645
- [Background] Akber A, Portale AA, Johansen KL. Use of pedometers to increase physical activity among children and adolescents with chronic kidney disease. Pediatr Nephrol. 2014 Aug;29(8):1395-402. doi: 10.1007/s00467-014-2787-6. Epub 2014 Mar 20. PMID 24648129
- [Background] Negri C, Bacchi E, Morgante S, Soave D, Marques A, Menghini E, Muggeo M, Bonora E, Moghetti P. Supervised walking groups to increase physical activity in type 2 diabetic patients. Diabetes Care. 2010 Nov;33(11):2333-5. doi: 10.2337/dc10-0877. PMID 20980426
- [Background] Applebaum MA, Lawson EF, von Scheven E. Perception of transition readiness and preferences for use of technology in transition programs: teens' ideas for the future. Int J Adolesc Med Health. 2013;25(2):119-25. doi: 10.1515/ijamh-2013-0019. PMID 23740658
- [Background] Ting TV, Kudalkar D, Nelson S, Cortina S, Pendl J, Budhani S, Neville J, Taylor J, Huggins J, Drotar D, Brunner HI. Usefulness of cellular text messaging for improving adherence among adolescents and young adults with systemic lupus erythematosus. J Rheumatol. 2012 Jan;39(1):174-9. doi: 10.3899/jrheum.110771. Epub 2011 Nov 15. PMID 22089460
- [Background] Takacs J, Pollock CL, Guenther JR, Bahar M, Napier C, Hunt MA. Validation of the Fitbit One activity monitor device during treadmill walking. J Sci Med Sport. 2014 Sep;17(5):496-500. doi: 10.1016/j.jsams.2013.10.241. Epub 2013 Oct 31. PMID 24268570
- [Background] James PA, Oparil S, Carter BL, Cushman WC, Dennison-Himmelfarb C, Handler J, Lackland DT, LeFevre ML, MacKenzie TD, Ogedegbe O, Smith SC Jr, Svetkey LP, Taler SJ, Townsend RR, Wright JT Jr, Narva AS, Ortiz E. 2014 evidence-based guideline for the management of high blood pressure in adults: report from the panel members appointed to the Eighth Joint National Committee (JNC 8). JAMA. 2014 Feb 5;311(5):507-20. doi: 10.1001/jama.2013.284427. PMID 24352797
- [Background] Tudor-Locke C, Pangrazi RP, Corbin CB, Rutherford WJ, Vincent SD, Raustorp A, Tomson LM, Cuddihy TF. BMI-referenced standards for recommended pedometer-determined steps/day in children. Prev Med. 2004 Jun;38(6):857-64. doi: 10.1016/j.ypmed.2003.12.018. PMID 15193909
- [Background] Pickering TG, Hall JE, Appel LJ, Falkner BE, Graves J, Hill MN, Jones DW, Kurtz T, Sheps SG, Roccella EJ. Recommendations for blood pressure measurement in humans and experimental animals: part 1: blood pressure measurement in humans: a statement for professionals from the Subcommittee of Professional and Public Education of the American Heart Association Council on High Blood Pressure Research. Circulation. 2005 Feb 8;111(5):697-716. doi: 10.1161/01.CIR.0000154900.76284.F6. PMID 15699287
- [Background] Flynn JT, Daniels SR, Hayman LL, Maahs DM, McCrindle BW, Mitsnefes M, Zachariah JP, Urbina EM; American Heart Association Atherosclerosis, Hypertension and Obesity in Youth Committee of the Council on Cardiovascular Disease in the Young. Update: ambulatory blood pressure monitoring in children and adolescents: a scientific statement from the American Heart Association. Hypertension. 2014 May;63(5):1116-35. doi: 10.1161/HYP.0000000000000007. Epub 2014 Mar 3. No abstract available. PMID 24591341
- [Derived] Bicki AC, Seth D, McCulloch CE, Lin F, Ku E. Use of activity trackers to improve blood pressure in young people at risk for cardiovascular disease: a pilot randomized controlled trial. Pediatr Nephrol. 2024 Aug;39(8):2467-2474. doi: 10.1007/s00467-024-06340-6. Epub 2024 Mar 19. PMID 38503990

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Six months of usual care without a device, followed by crossover to use of the physical activity tracker
- Physical Activity Tracker: FitBit: Daily use of physical activity tracker coupled with biweekly provider telemonitoring and feedback for 12 months
Period: Overall Study
Arm/Group | Usual Care | Physical Activity Tracker
Started | 21 | 42
Completed | 11 | 18
Not Completed | 10 | 24

BASELINE CHARACTERISTICS:
Groups:
- Usual Care Arm: Usual care x 6 months, then crossover to physical activity tracker x 6 months
- Intervention Arm: Physical activity tracker x 12 months
- Total: Total of all reporting groups
Arm/Group | Usual Care Arm | Intervention Arm | Total
Number analyzed (Participants) | 21 | 42 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.0 (4.4) | 17.6 (3.9) | 17.7 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 9 | 27 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 19 | 30
  Not Hispanic or Latino | 10 | 23 | 33
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 42 | 63
Estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73 m^2] | 81 (35) | 81 (25) | 81 (28)

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Office Systolic BP
Description: Change in mean systolic BP is modeled using all blood pressure data points collected between baseline and month 12 to provide an average change over time, accounting for repeated values from patients using a mixed linear regression approach.
Time Frame: Between baseline and month 12
Measure: Mean (95% Confidence Interval); unit: mmHg
Groups:
- Usual Care: Usual care x 6 months, then crossover to physical activity tracker x 6 months
- Physical Activity Tracker: Physical activity tracker x 12 months
Arm/Group | Usual Care | Physical Activity Tracker
Number analyzed (Participants) | 11 | 18
mmHg | 0.3 [-10 to 10] | -4 [-14 to 6]

2. Secondary Outcome: Number of Participants Retained
Description: Rate of study participant retention
Time Frame: Months 0-12
Measure: Count of Participants; unit: Participants
Groups:
- Usual Care Arm: Usual care for months 0-6, then crossover to use of physical activity tracker
- Intervention Arm: Use of physical activity tracker x 12 months
Arm/Group | Usual Care Arm | Intervention Arm
Number analyzed (Participants) | 21 | 42
Participants | 11 | 18

3. Secondary Outcome: Change in Weight (Z-score)
Description: Weights were measured in clinic using a standardized scale. Z score of 0 represents the population mean. A z-score of +1.96 represents the 95th percentile of weight and -1.96 represents the 5th percentile of weight. Change in weight (z-score) is modeled using all weight data points collected between baseline and month 12 to provide an average change over time accounting for repeated values from patients using a mixed linear regression approach.
Time Frame: Months 0-12
Measure: Mean (95% Confidence Interval); unit: Z-score
Arm/Group | Usual Care | Physical Activity Tracker
Number analyzed (Participants) | 11 | 18
Z-score | -0.20 [-0.34 to -0.07] | -0.06 [-0.17 to 0.05]

4. Primary Outcome: Change in Mean Office Systolic BP
Description: Change in mean systolic BP using blood pressure data points collected between baseline and month 6 to provide an average change over time
Time Frame: Between baseline and month 6
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Usual Care | Physical Activity Tracker
Number analyzed (Participants) | 18 | 26
mmHg | 3.0 [-2.5 to 8.4] | -2.3 [-6.5 to 1.8]

ADVERSE EVENTS:
Time Frame: Participants were followed during participation in the study for 1 year
Description: All-cause mortality Serious adverse events include hospitalizations related to the intervention and/or death
Groups:
- Usual Care Arm (mo. 0-6): Usual care for months 0-6
- Usual Care Arm (mo. 6-12): Crossover to use of physical activity tracker for control participants from months 6-12
Arm/Group | Usual Care Arm (mo. 0-6) | Usual Care Arm (mo. 6-12) | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/42
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT03325426/Prot_SAP_000.pdf